CLINICAL TRIAL: NCT01334931
Title: Preferential Use of Large Field of View During Image Acquisition for Coronary Angiography With Flat Detector Technology: a Simple Step to Reduce Radiation Exposure
Brief Title: Use of Large Field of View During Image Acquisition for Coronary Angiography
Acronym: XRay Reduction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Cristiano de Oliveira Cardoso, MD, MSc, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UP 4454/10
Record Dates: First submitted 2011-04-05; First posted 2011-04-13 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Exposure to Ionizing Radiation; Occupational Exposure to Radiation; Radiation Injury
Keywords: Exposure to Ionizing Radiation; Occupational Exposure to Radiation
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Large field of view (Experimental): Patients will have coronary angiography performed with large field of view lens
  Interventions: Radiation: Large field of view arm
- Medium field of view (Active Comparator): Patients will have coronary angiography performed with medium field of view lens
  Interventions: Radiation: Medium field of view

INTERVENTIONS:
Radiation: Large field of view arm — Patients will be allocated in the large field of view arm. Coronary angiography will be performed with large field of view lens (25 cm)
  Arms: Large field of view
Radiation: Medium field of view — Patients will be allocated in the medium field of view arm. Coronary angiography will be performed with medium field of view lens (20 cm)
  Arms: Medium field of view

SUMMARY:
Coronary angiography exposes patients and physicians to ionizing radiation. The purpose of this study is to evaluate the routine use of large field of view during image acquisition for coronary angiography. Patients with indication of diagnostic coronary angiography will be randomized for the use of either large field of view during image acquisition or medium field of view. Patients, physician and nurse radiation exposure will be measured by digital dosimeter.

ELIGIBILITY:
Inclusion Criteria:

* Indication of diagnostic coronary angiography for suspected coronary artery disease
* Sign written consent form

Exclusion Criteria:

* Therapeutics procedures
* Urgency/emergency procedures
* Previous CABG
* Severe valvular disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Patient's radiation exposure | 24 hours
  Patient's radiation exposure will be measured in mGy at the end of procedure

SECONDARY OUTCOMES:
Physician and nurse radiation exposure | 24 hours
  Physician and nurse radiation exposure will be measured in microSv at the end of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano O Cardoso, MD, MSc, Study Chair — Instituto de Cardiologia do Rio Grande do Sul
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil